CLINICAL TRIAL: NCT01120184
Title: A Randomized, 3 Arm, Multicenter, Phase III Study to Evaluate the Efficacy and the Safety of T-DM1 Combined With Pertuzumab or T-DM1 Combined With Pertuzumab-Placebo (Blinded for Pertuzumab), Versus the Combination of Trastuzumab Plus Taxane, as First Line Treatment in HER2 Positive Progressive or Recurrent Locally Advanced or Metastatic Breast Cancer
Brief Title: A Study of Trastuzumab Emtansine (T-DM1) Plus Pertuzumab/Pertuzumab Placebo Versus Trastuzumab [Herceptin] Plus a Taxane in Participants With Metastatic Breast Cancer (MARIANNE)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BO22589; 2009-017905-13 (EudraCT Number)
Record Dates: First submitted 2010-04-28; First posted 2010-05-10 (Estimated); Results first posted 2017-02-23 (Actual); Last update posted 2024-03-04 (Actual); Status verified 2024-02

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Docetaxel; Paclitaxel; pertuzumab; Trastuzumab; Ado-Trastuzumab Emtansine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Trastuzumab + Taxane (docetaxel or paclitaxel) (Experimental)
  Interventions: Drug: docetaxel; Drug: paclitaxel; Drug: trastuzumab [Herceptin]
- Trastuzumab emtansine + pertuzumab (Experimental)
  Interventions: Drug: pertuzumab; Drug: trastuzumab emtansine
- Trastuzumab emtansine + pertuzumab placebo (Experimental)
  Interventions: Drug: pertuzumab-placebo; Drug: trastuzumab emtansine

INTERVENTIONS:
Drug: docetaxel — 75 mg/m2 or 100 mg/m2 intravenously every 3 weeks for a minimum of 6 cycles.
  Arms: Trastuzumab + Taxane (docetaxel or paclitaxel)
Drug: paclitaxel — 80 mg/m2 intravenously weekly for a minimum of 18 weeks
  Arms: Trastuzumab + Taxane (docetaxel or paclitaxel)
Drug: pertuzumab — 840 mg intravenously on day 1 of cycle 1 followed by 420 mg intravenously every 3 weeks in subsequent cycles
  Arms: Trastuzumab emtansine + pertuzumab
Drug: pertuzumab-placebo — 840 mg intravenously on day 1 of cycle 1 followed by 420 mg intravenously every 3 weeks in subsequent cycles
  Arms: Trastuzumab emtansine + pertuzumab placebo
Drug: trastuzumab [Herceptin] — trastuzumab [Herceptin] doses when administered with docetaxel: 8 mg/kg intravenously on cycle 1 followed by 6 mg/kg every 3 weeks in subsequent cycles or trastuzumab (Herceptin) doses when administered with paclitaxel: 4 mg/kg intravenously on day 1 of cycle 1 followed by 2 mg/kg weekly starting on day 8 of cycle 1.
  Arms: Trastuzumab + Taxane (docetaxel or paclitaxel)
Drug: trastuzumab emtansine — 3.6 mg/kg intravenously every 3 weeks
  Arms: Trastuzumab emtansine + pertuzumab; Trastuzumab emtansine + pertuzumab placebo

SUMMARY:
This randomized, 3-arm, multicenter, phase III study will evaluate the efficacy and safety of trastuzumab emtansine (T-DM1) with pertuzumab or trastuzumab emtansine (T-DM1) with pertuzumab-placebo (blinded for pertuzumab), versus the combination of trastuzumab (Herceptin) plus taxane (docetaxel or paclitaxel) in participants with HER2-positive progressive or recurrent locally advanced or previously untreated metastatic breast cancer. Participants will be randomized to 1 of 3 treatment arms (Arms A, B or C). Arm A will be open-label, whereas Arms B and C will be blinded.

ELIGIBILITY:
Inclusion Criteria:

* Adult participants >/=18 years of age
* HER2-positive breast cancer
* Histologically or cytologically confirmed adenocarcinoma of the breast with locally recurrent or metastatic disease, and be a candidate for chemotherapy. Participants with locally advanced disease must have recurrent or progressive disease, which must not be amenable to resection with curative intent.
* Participants must have measurable and/or non-measurable disease which must be evaluable per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1
* Eastern Cooperative Oncology Group (ECOG) Performance Status 0 or 1
* Adequate organ function as determined by laboratory results

Exclusion Criteria:

* History of prior (or any) chemotherapy for metastatic breast cancer or recurrent locally advanced disease
* An interval of <6 months from the last dose of vinca-alkaloid or taxane cytotoxic chemotherapy until the time of metastatic diagnosis
* Hormone therapy <7 days prior to randomization
* Trastuzumab therapy and/or lapatinib (neo- or adjuvant setting) <21 days prior to randomization
* Prior trastuzumab emtansine or pertuzumab therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1095 (Actual)
Dates: Start 2010-07-31 (Actual); Primary Completion 2014-09-30 (Actual); Study Completion 2016-09-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (257):
- United States (62):
  - Uni of Arkansas For Medical Sciences; Arkansas Cancer Research Center, Little Rock, Arkansas
  - Scripps Cancer Center, La Jolla, California
  - University of California; Moores Cancer Center, La Jolla, California
  - Clnc L Trials & Rsch Assoc-Inc, Montebello, California
  - Southern California Kaiser Permanente, San Diego, California
  - Breastlink Medical Group Inc, Santa Ana, California
  - Kaiser Permanente; Oncology Clinical Trials, Vallejo, California
  - Smilow Cancer Hospital at Yale New Haven, New Haven, Connecticut
  - Innovative Medical Research of South Florida, Aventura, Florida
  - Northwest Oncology/ Hematology Assoc., Coral Springs, Florida
  - Florida Cancer Specialists; SCRI, Fort Myers, Florida
  - Mayo Clinic-Jacksonville, Jacksonville, Florida
  - Uni of Miami School of Medicine; Sylvester Comprehensive Cancer Center, Miami, Florida
  - University Cancer & Blood Center, LLC; Research, Athens, Georgia
  - Cancer Research Center of Hawaii; Clinical Sciences, Honolulu, Hawaii
  - Mountain States Tumor Inst., Boise, Idaho
  - Uni of Chicago, Chicago, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Ingalls Memorial Hospital, Harvey, Illinois
  - Loyola University Med Center, Maywood, Illinois
  - Illinois Cancer Care, Peoria, Illinois
  - Indiana University Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Horizon Oncology Research, Inc., Lafayette, Indiana
  - James Graham Brown Cancer Center, University of Louisville, Louisville, Kentucky
  - New England Cancer Specialists, Scarborough, Maine
  - Anne Arundel Health System Research Instit-Annapolis Oncology Ctr, Annapolis, Maryland
  - Boston Medical Center, Boston, Massachusetts
  - Spectrum Health Grand Rapids, Grand Rapids, Michigan
  - University of Minnesota., Minneapolis, Minnesota
  - Mayo Clinic Rochester, Rochester, Minnesota
  - Mercy Clinic Cancer & Hematology, Springfield, Missouri
  - St. John'S Mercy Medical Center; David C. Pratt Cancer Center, St Louis, Missouri
  - Dartmouth Hitchcock Med Center, Lebanon, New Hampshire
  - Hackensack Uni Medical Center; Northern Nj Cancer Center, Hackensack, New Jersey
  - Cancer Inst. of New Jersey, New Brunswick, New Jersey
  - San Juan Oncology Associates, Farmington, New Mexico
  - Queens Medical Associates, Fresh Meadows, New York
  - Queens Hospital Center, Jamaica, New York
  - Arena Oncology Associates, Lake Success, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Weill Medical College of Cornell Uni, New York, New York
  - Carolinas Hem-Oncology Assoc, Charlotte, North Carolina
  - Carolina Oncology Specialists, PA - Hickory, Hickory, North Carolina
  - Marion L. Shepard Cancer Center, Washington, North Carolina
  - Sanford Roger Maris Cancer Center, Fargo, North Dakota
  - Oncology Hematology Care - SCRI, Cincinnati, Ohio
  - Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Charleston Oncology, P .A, Charleston, South Carolina
  - Medical University of SC (MUSC), Charleston, South Carolina
  - South Carolina Oncology Associates - SCRI, Columbia, South Carolina
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - SCRI Tennessee Oncology Chattanooga, Chattanooga, Tennessee
  - West Clinic, Germantown, Tennessee
  - Tennessee Onc., PLLC - SCRI, Nashville, Tennessee
  - Vanderbilt-Ingram Cancer Ctr, Nashville, Tennessee
  - The Don & Sybil Harrington Cancer Center; Department of Clinical Research, Amarillo, Texas
  - Uni of Texas Southwestern Medical Center, Dallas, Texas
  - Uni of Texas - Md Anderson Cancer Center; Dept of Breast Medical Oncology, Houston, Texas
  - Northern Utah Associates, Ogden, Utah
  - The Providence Regional Medical Center Everett, Everett, Washington
  - University of Washington, Seattle, Washington
  - Northwest Medical Specialties, Tacoma, Washington
- Argentina (2):
  - Fundación Investigar, Buenos Aires
  - Centro Medico San Roque, San Miguel de Tucumán
- Australia (5):
  - Mater Misericordiae Hospital; Chemotherapy Cottage, Sydney, New South Wales
  - Calvary Mater Newcastle; Medical Oncology, Waratah, New South Wales
  - Wesley Medical Centre; Clinic For Haematology and Oncology, Auchenflower, Queensland
  - Royal Adelaide Hospital; Oncology, Adelaide, South Australia
  - Peter Maccallum Cancer Institute; Medical Oncology, Melbourne, Victoria
- Austria (2):
  - Lkh Salzburg - Univ. Klinikum Salzburg; Iii. Medizinische Abt., Salzburg
  - Medizinische Universität Wien; Univ.Klinik für Innere Medizin I - Abt. für Onkologie, Vienna
- Belgium (3):
  - Cliniques Universitaires St-Luc, Brussels
  - Clinique Ste-Elisabeth, Namur
  - Sint Augustinus Wilrijk, Wilrijk
- Bosnia and Herzegovina (2):
  - University Clinical Centre of the Republic of Srpska, Banja Luka
  - Clinic of Oncology, University Clinical Center Sarajevo, Sarajevo
- Brazil (8):
  - *X*Instituto Nacional do Cancer - INCA, Rio de Janeiro, Rio de Janeiro
  - Liga Norte Riograndense Contra O Câncer, Natal, Rio Grande do Norte
  - Hospital Nossa Senhora da Conceicao, Porto Alegre, Rio Grande do Sul
  - Clinica de Oncologia de Porto Alegre - CliniOnco, Porto Alegre, Rio Grande do Sul
  - Hospital Sao Lucas - PUCRS, Porto Alegre, Rio Grande do Sul
  - Clinica de Neoplasias Litoral, Itajaí, Santa Catarina
  - Instituto do Cancer do Estado de Sao Paulo - ICESP, São Paulo, São Paulo
  - Hospital Perola Byington, São Paulo, São Paulo
- Canada (4):
  - Cross Cancer Institute; Clinical Trials, Edmonton, Alberta
  - North York General Hospital, Toronto, Ontario
  - Cuse - Centre Universitaire De Sante; Site Fleurimont, Sherbrooke, Quebec
  - CHU de Québec ? Hôpital du Saint-Sacrement / ONCOLOGY, Québec
- Colombia (4):
  - Clinica del Country, Bogotá
  - Instituto Colombiano Para El Avance De La Medicina: Icamedic, Bucaramanga
  - Centro Medico Imbanaco, Cali
  - Instituto Cancerologico de Nariño, Pasto
- Czechia (4):
  - Masarykuv onkologicky ustav, Brno
  - Fakultni nemocnice Olomouc; Onkologicka klinika, Olomouc
  - Fakultni Poliklinika Vseobecne Fakultni Niemocnice; Onkologicka Klinika, Prague
  - Fakultni Nemocnice Na Bulovce; Ustav Radiacni Onkologie, Prague
- Vejle Sygehus; Onkologisk Afdeling, Vejle, Denmark
- France (12):
  - HOPITAL JEAN MINJOZ; Oncologie, Besançon
  - Centre Jean Perrin; Hopital De Jour, Clermont-Ferrand
  - Centre Oscar Lambret; Senologie, Lille
  - Institut Paoli Calmettes; Oncologie Medicale, Marseille
  - Institut régional du Cancer Montpellier, Montpellier
  - Centre D'Oncologie de Gentilly; Oncology, Nancy
  - Institut Curie; Oncologie Medicale, Paris
  - Hopital Saint Louis; Service Onco Thoracique, Paris
  - HOPITAL TENON; Cancerologie Medicale, Paris
  - Chu La Miletrie; Radiotherapie, Poitiers
  - Centre Rene Huguenin; ONCOLOGIE GENETIQUE, Saint-Cloud
  - Institut de Cancerologie de La Loire; Radiotherapie, Saint-Priest-en-Jarez
- Germany (10):
  - Klinikum Essen-Mitte Ev. Huyssens-Stiftung / Knappschafts GmbH; Klinik für Senologie / Brustzentrum, Essen
  - Universitätsklinikum Halle (Saale); Universitätsklinik Und Poliklinik Für Gynäkologie, Halle
  - Facharztzentrum Eppendorf, Studien GbR, Hamburg
  - MVZ Onko Medical GmbH Hannover, Ralf Lohse (Geschäftsführer), Hanover
  - Nationales Centrum für Tumorerkrankungen (NCT) ; Gyn. Onk. Frauenklinik; Uniklinikum Heidelberg, Heidelberg
  - Universitätsklinikum Magdeburg; Frauenheilkunde & Geburtshilfe, Magdeburg
  - Universitätsmedizin Mainz; Klinik u. Poliklinik f. Geburtshilfe u. Frauenheilkunde, Mainz
  - Mühlenkreiskliniken; Johannes Wesling Klinikum Minden; Klinik für Frauenheilkunde und Geburtshilfe, Minden
  - Rotkreuzklinikum München; Frauenklinik, München
  - Klinikum Mutterhaus der Borromaeerinnen gGmbH; Haematologie/Onkologie, Trier
- Greece (3):
  - Alexandras General Hospital of Athens; Oncology Department, Athens
  - Univ General Hosp Heraklion; Medical Oncology, Heraklion
  - University Hospital of Larissa; Oncology, Larissa
- Guatemala (2):
  - Centro Oncológico Sixtino / Centro Oncológico SA, Guatemala City
  - Grupo Angeles, Guatemala City
- Hungary (4):
  - Szent Margit Hospital; Dept. of Oncology, Budapest
  - Semmelweis Egyetem Onkologiai Központ, Budapest
  - Semmelweis Egyetem Aok; Iii.Sz. Belgyogyaszati Klinika, Budapest
  - Pécsi Tudományegyetem; Klinikai Központ Onkoterápiás Intézet, Pécs
- Italy (13):
  - Campus Universitario S.Venuta; Centro Oncologico T.Campanella, Catanzaro, Calabria
  - IRST Istituto Scientifico Romagnolo Per Lo Studio E Cura Dei Tumori, Sede Meldola; Oncologia Medica, Meldola, Emilia-Romagna
  - A.O. Universitaria Policlinico Di Modena; Ematologia, Modena, Emilia-Romagna
  - Arcispedale Santa Maria Nuova; Oncologia, Reggio Emilia, Emilia-Romagna
  - Ospedale Degli Infermi; Divisione Di Oncologia, Rimini, Emilia-Romagna
  - Azienda Ospedaliero-Universitaria Dipartimento Interaziendale Di Oncologia, Udine, Friuli Venezia Giulia
  - Istituto Europeo Di Oncologia, Milan, Lombardy
  - Fondazione Salvatore Maugeri, Pavia, Lombardy
  - IRCCS Istituto Clinico Humanitas; Oncologia, Rozzano (MI), Lombardy
  - Centro Catanese Di Oncologia; Oncologia Medica, Catania, Sicily
  - Ospedale Papardo- Piemonte;Oncologia Medica, Messina, Sicily
  - Ospedale Misericordia E Dolce; Oncologia Medica, Prato, Tuscany
  - Azienda Ospedaliera Di Perugia Ospedale s. Maria Della Misericordia; Oncologia Medica, Perugia, Umbria
- Japan (28):
  - Aichi Cancer Center Hospital, Breast Oncology, Aichi
  - Natl Hosp Org Shikoku; Cancer Ctr, Surgery, Ehime
  - National Hospital Organization Kyushu Cancer Center;Breast Oncology, Fukuoka
  - Gifu University Hospital; Digestive Surgery, Gifu
  - Hiroshima University Hospital; Breast Surgery, Hiroshima
  - National Hospital Organization Hokkaido Cancer Center; Breast Surgery, Hokkaido
  - Hyogo College Of Medicine; Breast And Endocrine Surgery, Hyōgo
  - Hyogo Cancer Center; Breast Surgery, Hyōgo
  - Kanazawa University Hospital; Breast Oncology, Ishikawa
  - Sagara Hospital; Breast Surgery, Kagoshima
  - Tokai University Hospital, Breast Surgery, Kanagawa
  - Kumamoto University Hospital; Breast and Endocrine Surgery, Kumamoto
  - Kumamoto City Hospital, Breast and Endocrine Surgery, Kumamoto
  - Kyoto University Hospital; Breast Surgery, Kyoto
  - Tohoku University Hospital; General Surgery, Miyagi
  - Niigata Cancer Ctr Hospital; Breast Surgery, Niigata
  - Iwate Med Univ School of Med; Surgery, Numakunai
  - Kawasaki Medical School Hospital; Breast and Thyroid Surgery, Okayama
  - National Hospital Organization Osaka National Hospital; Breast Surgery, Osaka
  - Osaka University Hospital; Breast and Endocrine Surgery, Osaka
  - Saitama Medical University International Medical Center; Medical Oncology, Saitama
  - Saitama Cancer Center, Breast Oncology, Saitama
  - Shizuoka Cancer Center; Breast Surgery, Shizuoka
  - Shizuoka General Hospital; Breast Surgery, Shizuoka
  - National Cancer Center Hospital; Medical Oncology, Tokyo
  - Toranomon Hospital; Breast and Endocrine Surgery, Tokyo
  - The Cancer Inst. Hosp. of JFCR; Breast Oncology Center, Tokyo
  - Tokyo Medical Uni. Hospital; Breast Oncology, Tokyo
- Malaysia (3):
  - Pantai Hospital Kuala Lumpur; Dept of Oncology & Radiotherapy, Kuala Lumpur, FED. Territory of Kuala Lumpur
  - Sunway Medical Centre, Kuala Selangor, Selangor
  - Beacon International Specialist Centre, Petaling Jaya, Selangor, Selangor
- Mexico (6):
  - Centro de Investigacion; Clinica Del Pacifico, Acapulco de Juárez, Guerrero
  - Centro Universitario Contra El Cancer, Monterrey, Nuevo León
  - Oaxaca Site Management Organization, Oaxaca City, Oaxaca
  - Hospital Privado San Jose; Oncologia, Obregón, Sonora
  - Centenario Hospital Miguel Hidalgo, Aguascalientes
  - Centro Oncológico Estatal; ISSSEMYM Oncología, Toluca
- New Zealand (2):
  - Auckland city hospital; Auckland Regional Cancer Centre and Blood Service, Auckland
  - Waikato Hospital; Regional Cancer Center, Hamilton
- Private Health Organization Acibadem Sistina Hospital, Skopje, North Macedonia
- The Panama Clinic, Panama City, Panama
- Peru (3):
  - Hospital Nacional Carlos Alberto Seguin Escobedo-Essalud; Oncology & Haemathology, Arequipa
  - Hospital Nacional Edgardo Rebagliati Martins; Oncologia, Lima
  - Unidad de Investigacion Oncologia Clinica ? Piura; Unidad de Oncología Clínica, Piura
- Philippines (2):
  - Cebu Cancer Institute; Perpetual Succour Hospital, Cebu City
  - Cardinal Santos Medical Center, San Juan City
- Poland (5):
  - Centrum Onkologii;Im. Franciszka Lukaszczyka;Onkologii, Bydgoszcz
  - Medical University of Gdansk, Gdansk
  - Centrum Onkologii, Instytut, Klinika Chemioterapii; Oddzial Chemoterapii, Krakow
  - COZL Oddzial Onkologii Klinicznej z pododdzialem Chemioterapii Dziennej, Lublin
  - Cent.Onkologii-Instytut im. M. S-Curie, Klinika Now. Piersi i Chirurgii Rekon, Warsaw
- IPO do Porto; Servico de Oncologia Medica, Porto, Portugal
- Romania (3):
  - Coltea Hospital; Oncology, Bucharest
  - Cluj Clinical County Hospital; Oncology Dept, Cluj-Napoca
  - Prof. Dr. I. Chiricuta Institute of Oncology, Cluj-Napoca
- Russia (10):
  - Moscow city oncology hospital; #62 of Moscow Healthcare Department, Moscow, Moscow Oblast
  - Blokhin Cancer Research Center; Combined Treatment, Moskva, Moscow Oblast
  - Ryazan State Medical University Named after I.P.Pavlov, Ryazan, Ryazan Oblast
  - State Budget Institution of Healthcare of Stavropol region Pyatigorsk Oncology Dispensary, Pyatigorsk, Stavropol Kray
  - Clinical Oncology Dispensary of Ministry of Health of Tatarstan, Kazan', Tatarstan Republic
  - Ivanovo Regional Oncology Dispensary, Ivanovo
  - SBI of Healthcare Samara Regional Clinical Oncology Dispensary, Samara
  - SBI of Healthcare of Stavropol region Stavropol Regional Clinical Oncology Dispensary, Stavropol
  - Tula Regional Oncology Dispensary, Tula
  - GUZ Vladimir Regional Clinical Oncological Dispensary, Vladimir
- South Korea (5):
  - Seoul National University Bundang Hospital; Hematology Medical Oncology, Gyeonggi-do
  - Seoul National Uni Hospital; Dept. of Internal Medicine/Hematology/Oncology, Seoul
  - Samsung Medical Centre; Division of Hematology/Oncology, Seoul
  - Asan Medical Center, Uni Ulsan Collegemedicine; Dept.Internal Medicine / Divisionhematology/Oncology, Seoul
  - Korea University Guro Hospital; Oncology, Seoul
- Spain (11):
  - Hospital General Universitario de Elche; Servicio de Oncologia, Elche, Alicante
  - Hospital Univ Vall d'Hebron; Servicio de Oncologia, Sant Andreu de la Barca, Barcelona
  - Complejo Hospitalario Universitario de Santiago (CHUS) ; Servicio de Oncologia, Santiago de Compostela, LA Coruña
  - Complejo Hospitalario Universitario A Coruña (CHUAC, Materno Infantil), Oncología, A Coruña
  - Hospital del Mar; Servicio de Oncologia, Barcelona
  - Complejo Hospitalario de Jaen-Hospital Universitario Medico Quirurgico; Servicio de Oncologia, Jaén
  - Hospital General Universitario Gregorio Marañon; Servicio de Oncologia, Madrid
  - Hospital Universitario 12 de Octubre; Servicio de Oncologia, Madrid
  - Hospital Universitario La Paz; Servicio de Oncologia, Madrid
  - Hospital Clinico Universitario Virgen de la Victoria; Servicio de Oncologia, Málaga
  - Hospital Clinico Universitario de Valencia; Servicio de Onco-hematologia, Valencia
- Skånes Universitetssjukhus; Kliniska Forskningsenheten Onkologimottagning medicinsk behandling, Malmo, Sweden
- Switzerland (3):
  - Kantonsspital Baden; Medizinische Klinik, Onkologie, Baden
  - Universitaetsspital Basel; Onkologie, Basel
  - Kantonsspital Graubünden Medizin Onkologie; Onkologie und Hämatologie, Chur
- Taiwan (4):
  - Changhua Christian Hospital; Hematology-Oncology, Changhua
  - Kaohsiung Medical Uni Chung-Ho Hospital; Dept of Surgery, Kaohsiung City
  - National Taiwan Uni Hospital; Dept of Oncology, Taipei
  - Tri-Service General Hospital; Hematology and Oncology, Taipei
- Thailand (6):
  - National Cancer Inst., Bangkok
  - Rajavithi Hospital; Division of Medical Oncology, Bangkok
  - Ramathibodi Hospital; Dept of Med.-Div. of Med. Onc, Bangkok
  - Faculty of Med. Siriraj Hosp.; Med.-Div. of Med. Oncology, Bangkok
  - Maharaj Nakorn Hospital; Internal Medicine, Chiang Mai
  - Songklanagarind Hospital; Department of Oncology, Songkhla
- Oncology Consultants Limited, Nassau, The Bahamas
- Turkey (Türkiye) (4):
  - Baskent University Adana Dr. Turgut Noyan Practice and Research Hospital; Medical Oncology, Adana
  - Cukurova Uni Faculty of Medicine; Medical Oncology, Adana
  - Gazi Uni Medical Faculty Hospital; Oncology Dept, Ankara
  - Ege Uni Medical Faculty Hospital; Oncology Dept, Izmir
- United Kingdom (16):
  - Bristol Haematology and Oncology centre, Bristol
  - Cambridge University Hospitals NHS Foundation Trust, Cambridge
  - Royal Cornwall Hospital; Dept of Clinical Oncology, Cornwall
  - The Beatson West of Scotland Cancer Centre; Cancer Clinical Trials Unit, Glasgow
  - Leicester Royal Infirmary; Dept. of Medical Oncology, Leicester
  - Royal Free Hospital; Dept of Oncology, London
  - Guys Hospital; Management Offices, London
  - Royal Marsden Hospital; Dept of Med-Onc, London
  - Christie Hospital; Breast Cancer Research Office, Manchester
  - Nottingham City Hospital; Oncology, Nottingham
  - Peterborough City Hospital; Oncology Ward, Peterborough
  - Queen Alexandra Hospital, Portsmouth, Portsmouth
  - Weston Park Hospital; Cancer Clinical Trials Centre, Sheffield
  - Southampton General Hospital; Somers Cancer Research Building, Southampton
  - Uni Hospital of North Staffordshire; Staffordshire Oncology Centre, Stoke-on-Trent
  - Royal Marsden Hospital; Dept of Medical Oncology, Sutton

REFERENCES:
- [Derived] Perez EA, de Haas SL, Eiermann W, Barrios CH, Toi M, Im YH, Conte PF, Martin M, Pienkowski T, Pivot XB, Burris HA 3rd, Stanzel S, Patre M, Ellis PA. Relationship between tumor biomarkers and efficacy in MARIANNE, a phase III study of trastuzumab emtansine +/- pertuzumab versus trastuzumab plus taxane in HER2-positive advanced breast cancer. BMC Cancer. 2019 May 30;19(1):517. doi: 10.1186/s12885-019-5687-0. PMID 31146717
- [Derived] Bighin C, Pronzato P, Del Mastro L. Trastuzumab emtansine in the treatment of HER-2-positive metastatic breast cancer patients. Future Oncol. 2013 Jul;9(7):955-7. doi: 10.2217/fon.13.74. PMID 23837759
- [Derived] Scott AM, Wolchok JD, Old LJ. Antibody therapy of cancer. Nat Rev Cancer. 2012 Mar 22;12(4):278-87. doi: 10.1038/nrc3236. PMID 22437872

RESULTS

PARTICIPANT FLOW:
Groups:
- Trastuzumab + Taxane: Participants received trastuzumab plus either docetaxel or paclitaxel. The regimen was chosen at the investigator's discretion. Option 1: trastuzumab 8 mg/kg via IV infusion on Day 1 of Cycle 1, then 6 mg/kg IV on Day 1 of each subsequent 3-week cycle; plus a minimum of 6 cycles with docetaxel 75 or 100 mg/m^2 IV on Day 1 of each 3-week cycle. Option 2: trastuzumab 4 mg/kg IV on Day 1 of Cycle 1, then 2 mg/kg IV weekly beginning on Day 8 of Cycle 1; plus a minimum of 18 weeks with paclitaxel 80 mg/m^2 IV weekly. Treatment continued until disease progression, unacceptable toxicity, or study termination. If trastuzumab or docetaxel were discontinued for toxicity, the other agent could be continued as monotherapy.
- Trastuzumab Emtansine + Placebo: Participants received trastuzumab emtansine plus pertuzumab-placebo. Trastuzumab emtansine was administered as 3.6 mg/kg via IV infusion, following completion of the placebo IV infusion, on Day 1 of each 3-week cycle. Treatment continued until disease progression, unacceptable toxicity, or study termination.
- Trastuzumab Emtansine + Pertuzumab: Participants received trastuzumab emtansine plus pertuzumab. Trastuzumab emtansine was administered as 3.6 mg/kg via IV infusion, following completion of the pertuzumab IV infusion, on Day 1 of each 3-week cycle. Pertuzumab was given as 840 mg IV on Day 1 of Cycle 1, then 420 mg IV on Day 1 of each subsequent 3-week cycle. Treatment continued until disease progression, unacceptable toxicity, or study termination.
Period: Overall Study
Arm/Group | Trastuzumab + Taxane | Trastuzumab Emtansine + Placebo | Trastuzumab Emtansine + Pertuzumab
Started | 365 | 367 | 363
Treated | 355 | 365 | 360
Completed | 0 | 0 | 0
Not Completed | 365 | 367 | 363
Not completed — Adverse Event | 0 | 1 | 0
Not completed — Lost to Follow-up | 13 | 13 | 11
Not completed — Physician Decision | 9 | 1 | 3
Not completed — Reason not Specified | 8 | 3 | 12
Not completed — Sponsor Decision to Terminate Study | 133 | 144 | 143
Not completed — Subject/ Guardian Decision to Withdraw | 32 | 29 | 25
Not completed — Death | 170 | 176 | 169

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat (ITT) Population: All participants randomized in the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Trastuzumab + Taxane | Trastuzumab Emtansine + Placebo | Trastuzumab Emtansine + Pertuzumab | Total
Number analyzed (Participants) | 365 | 367 | 363 | 1095
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.2 (11.3) | 52.6 (11.4) | 52.2 (12.0) | 53.0 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 362 | 365 | 361 | 1088
  Male | 3 | 2 | 2 | 7

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Death or Disease Progression According to Independent Review Facility (IRF) Assessment
Description: Tumor assessments were performed according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1, using radiographic images submitted to the IRF up to and including the confirmatory tumor assessment 4 to 6 weeks after study drug discontinuation. Disease progression was defined as a greater than or equal to (≥) 20 percent (%) and 5-millimeter (mm) increase in sum of diameters of target lesions, taking as reference the smallest sum obtained during the study, or appearance of new lesion(s). The percentage of participants with death or disease progression was calculated as [number of participants with event divided by the number analyzed] multiplied by 100.
Time Frame: Up to 48 months from randomization until clinical cutoff of 16-Sept-2014 (at Screening, every 9 weeks for 81 weeks, then every 12 weeks thereafter and/or up to 42 days after last dose)
Population: ITT Population.
Measure: Number; unit: percentage of participants
Arm/Group | Trastuzumab + Taxane | Trastuzumab Emtansine + Placebo | Trastuzumab Emtansine + Pertuzumab
Number analyzed (Participants) | 365 | 367 | 363
percentage of participants | 63.3 | 64.3 | 59.8

2. Primary Outcome: Progression-Free Survival (PFS) According to IRF Assessment
Description: Tumor assessments were performed according to RECIST version 1.1, using radiographic images submitted to the IRF up to and including the confirmatory tumor assessment 4 to 6 weeks after study drug discontinuation. PFS was defined as the time from randomization to first documented disease progression or death from any cause. Disease progression was defined as a ≥20% and 5-mm increase in sum of diameters of target lesions, taking as reference the smallest sum obtained during the study, or appearance of new lesion(s). Median duration of PFS was estimated using Kaplan-Meier analysis, and corresponding confidence intervals (CIs) were computed using the Brookmeyer-Crowley method.
Time Frame: as for outcome 1
Population: ITT Population.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Trastuzumab + Taxane | Trastuzumab Emtansine + Placebo | Trastuzumab Emtansine + Pertuzumab
Number analyzed (Participants) | 365 | 367 | 363
months | 13.7 [12.4 to 14.9] | 14.1 [10.9 to 16.8] | 15.2 [12.5 to 18.8]
Statistical Analysis 1: Comparison: Trastuzumab + Taxane vs Trastuzumab Emtansine + Placebo; Stratified Analysis: Stratification factors included world region (United States, Western Europe/Canada/Australia-Pacific, Eastern Europe, Asia, others); prior adjuvant/neoadjuvant therapy (no, yes [trastuzumab and/or lapatinib], yes [no trastuzumab and/or lapatinib]), and visceral disease (present, absent); Test type: Non-Inferiority or Equivalence — The study was powered for superiority with target hazard ratio (HR) equal to 0.75, as well as for non-inferiority with HR equal to 1.1765 for comparison between each of the trastuzumab emtansine-containing arms and the trastuzumab + taxane arm. Non-inferiority was established if the upper bound of the 97.5% CI was less than (<) 1.1765. Superiority was achieved if the upper bound of the 97.5% CI was <1.00; p = 0.3125, Log Rank — Test and p-value apply for superiority test. Two-sided significance level of 2.5% was used to adjust for independent comparison between each of the trastuzumab emtansine-containing arms and the trastuzumab + taxane arm; Hazard Ratio (HR) = 0.91, 97.5% CI 2-sided [0.73 to 1.13] — Direction of comparison: Trastuzumab Emtansine + Placebo vs. Trastuzumab + Taxane
Statistical Analysis 2: Comparison: Trastuzumab + Taxane vs Trastuzumab Emtansine + Pertuzumab; [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority or Equivalence — The study was powered for superiority with target HR equal to 0.75, as well as for non-inferiority with HR equal to 1.1765 for comparison between each of the trastuzumab emtansine-containing arms and the trastuzumab + taxane arm. Non-inferiority was established if the upper bound of the 97.5% CI was <1.1765. Superiority was achieved if the upper bound of the 97.5% CI was <1.00; p = 0.1407, Log Rank — [p-value comment as in outcome 2, analysis 1]; Hazard Ratio (HR) = 0.87, 97.5% CI 2-sided [0.69 to 1.08] — Direction of comparison: Trastuzumab Emtansine + Pertuzumab vs. Trastuzumab + Taxane
Statistical Analysis 3: Comparison: Trastuzumab Emtansine + Placebo vs Trastuzumab Emtansine + Pertuzumab; [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority or Equivalence — The study was powered for superiority with target HR equal to 0.75, as well as for non-inferiority with HR equal to 1.1765 for comparison between each of the trastuzumab emtansine-containing arms and the trastuzumab + taxane arm; p = 0.3075, Log Rank — Test and p-value apply for superiority test. Primary endpoint did not meet superiority of PFS for trastuzumab emtansine + pertuzumab versus trastuzumab + taxane (two-sided significance level 2.5%); thus, tests and p-value are considered descriptive; Hazard Ratio (HR) = 0.91, 97.5% CI 2-sided [0.73 to 1.13] — Direction of comparison: Trastuzumab Emtansine + Pertuzumab vs. Trastuzumab Emtansine + Placebo

3. Secondary Outcome: Percentage of Participants Who Died Prior to Clinical Cutoff
Description: The percentage of participants who died prior to clinical cutoff was calculated as [number of participants with event divided by the number analyzed] multiplied by 100.
Time Frame: Up to 70 months from randomization until clinical cutoff of 15-May-2016 (every 3 months until death, loss to follow-up, withdrawal, or study termination)
Population: ITT Population.
Measure: Number; unit: percentage of participants
Arm/Group | Trastuzumab + Taxane | Trastuzumab Emtansine + Placebo | Trastuzumab Emtansine + Pertuzumab
Number analyzed (Participants) | 365 | 367 | 363
percentage of participants | 46.3 | 47.7 | 46.3

4. Secondary Outcome: Overall Survival (OS) at Clinical Cutoff
Description: OS was defined as the time from randomization to death from any cause. Median duration of OS was estimated using Kaplan-Meier analysis, and corresponding CIs were computed using the Brookmeyer-Crowley method.
Time Frame: as for outcome 3
Population: ITT Population.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Trastuzumab + Taxane | Trastuzumab Emtansine + Placebo | Trastuzumab Emtansine + Pertuzumab
Number analyzed (Participants) | 365 | 367 | 363
months | 50.86 [44.75 to 60.75] | 53.68 [48.36 to 64.36] | 51.78 [47.87 to NA] — Upper limit of CI was not reached due to low number of participants with events.
Statistical Analysis 1: Comparison: Trastuzumab + Taxane vs Trastuzumab Emtansine + Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.6568, Log Rank; Hazard Ratio (HR) = 0.93, 97.5% CI 2-sided [0.73 to 1.20] — Direction of comparison: Trastuzumab Emtansine + Placebo vs Trastuzumab + Taxane
Statistical Analysis 2: Comparison: Trastuzumab + Taxane vs Trastuzumab Emtansine + Pertuzumab; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.5691, Log Rank; Hazard Ratio (HR) = 0.86, 97.5% CI 2-sided [0.67 to 1.11] — Direction of comparison: Trastuzumab Emtansine + Pertuzumab vs Trastuzumab + Taxane

5. Secondary Outcome: Percentage of Participants With Death or Disease Progression According to Investigator Assessment
Description: Tumor assessments were performed by the investigator according to RECIST version 1.1. Disease progression was defined as a ≥20% and 5-mm increase in sum of diameters of target lesions, taking as reference the smallest sum obtained during the study, or appearance of new lesion(s). The percentage of participants with death or disease progression was calculated as [number of participants with event divided by the number analyzed] multiplied by 100.
Time Frame: as for outcome 1
Population: ITT Population.
Measure: Number; unit: percentage of participants
Arm/Group | Trastuzumab + Taxane | Trastuzumab Emtansine + Placebo | Trastuzumab Emtansine + Pertuzumab
Number analyzed (Participants) | 365 | 367 | 363
percentage of participants | 72.1 | 70.3 | 67.5

6. Secondary Outcome: PFS According to Investigator Assessment
Description: Tumor assessments were performed by the investigator according to RECIST version 1.1. PFS was defined as the time from randomization to first documented disease progression or death from any cause. Disease progression was defined as a ≥20% and 5-mm increase in sum of diameters of target lesions, taking as reference the smallest sum obtained during the study, or appearance of new lesion(s). Median duration of PFS was estimated using Kaplan-Meier analysis, and corresponding CIs were computed using the Brookmeyer-Crowley method.
Time Frame: as for outcome 1
Population: ITT Population.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Trastuzumab + Taxane | Trastuzumab Emtansine + Placebo | Trastuzumab Emtansine + Pertuzumab
Number analyzed (Participants) | 365 | 367 | 363
months | 12.5 [10.5 to 13.6] | 14.1 [12.2 to 16.7] | 14.8 [12.4 to 17.8]
Statistical Analysis 1: Comparison: Trastuzumab + Taxane vs Trastuzumab Emtansine + Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; Hazard Ratio (HR) = 0.85, 97.5% CI 2-sided [0.69 to 1.04] — Direction of comparison: Trastuzumab Emtasine + Placebo vs Trastuzumab + Taxane
Statistical Analysis 2: Comparison: Trastuzumab + Taxane vs Trastuzumab Emtansine + Pertuzumab; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; Hazard Ratio (HR) = 0.77, 97.5% CI 2-sided [0.63 to 0.95] — Direction of comparison: Trastuzumab Emtansine + Pertuzumab vs Trastuzumab + Taxane

7. Secondary Outcome: Percentage of Participants Experiencing Treatment Failure
Description: Treatment failure was defined as the discontinuation of all study medications in the treatment arm for any reason including disease progression, treatment toxicity, death, physician decision, or participant withdrawal. The percentage of participants with treatment failure was calculated as [number of participants with event divided by the number analyzed] multiplied by 100.
Time Frame: Up to 48 months from randomization until clinical cutoff of 16-Sept-2014
Population: ITT Population.
Measure: Number; unit: percentage of participants
Arm/Group | Trastuzumab + Taxane | Trastuzumab Emtansine + Placebo | Trastuzumab Emtansine + Pertuzumab
Number analyzed (Participants) | 365 | 367 | 363
percentage of participants | 85.8 | 82.6 | 80.2

8. Secondary Outcome: Time to Treatment Failure (TTF)
Description: Treatment failure was defined as the discontinuation of all study medications in the treatment arm for any reason including disease progression, treatment toxicity, death, physician decision, or participant withdrawal. TTF was defined as the time from randomization to treatment failure. Median TTF was estimated using Kaplan-Meier analysis, and corresponding CIs were computed using the Brookmeyer-Crowley method.
Time Frame: Up to 48 months from randomization until clinical cutoff of 16-Sept-2014
Population: ITT Population.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Trastuzumab + Taxane | Trastuzumab Emtansine + Placebo | Trastuzumab Emtansine + Pertuzumab
Number analyzed (Participants) | 365 | 367 | 363
months | 10.2 [9.2 to 11.8] | 12.1 [9.9 to 13.9] | 11.8 [9.9 to 14.2]
Statistical Analysis 1: Comparison: Trastuzumab + Taxane vs Trastuzumab Emtansine + Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; Hazard Ratio (HR) = 0.80, 97.5% CI 2-sided [0.66 to 0.97] — Direction of comparison: Trastuzumab Emtansine + Placebo vs Trastuzumab + Taxane
Statistical Analysis 2: Comparison: Trastuzumab + Taxane vs Trastuzumab Emtansine + Pertuzumab; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; Hazard Ratio (HR) = 0.78, 97.5% CI 2-sided [0.65 to 0.95] — Direction of comparison: Trastuzumab Emtansine + Pertuzumab vs Trastuzumab + Taxane

9. Secondary Outcome: One-Year Survival Rate
Description: The percentage of participants alive at 1 year after randomization was estimated as the one-year survival rate using Kaplan-Meier analysis, and corresponding CIs were computed using Greenwood's estimate of the standard error.
Time Frame: From randomization until 1 year
Population: ITT Population.
Measure: Number (95% Confidence Interval); unit: percentage probability of being alive
Arm/Group | Trastuzumab + Taxane | Trastuzumab Emtansine + Placebo | Trastuzumab Emtansine + Pertuzumab
Number analyzed (Participants) | 365 | 367 | 363
percentage probability of being alive | 91.4 [88.44 to 94.41] | 92.4 [89.62 to 95.15] | 91.9 [89.00 to 94.77]

10. Secondary Outcome: Percentage of Participants With Grade ≥3 Adverse Events
Description: Adverse events were graded according to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.0. Grade 3: Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self care activity of daily living with inability to perform bathing, dressing and undressing, feeding self, using the toilet, taking medications but not bedridden. Grade 4: An immediate threat to life. Urgent medical intervention is required in order to maintain survival. Grade 5: Death.
Time Frame: Up to 50 months from randomization until clinical cutoff of 16-Sept-2014 (continuously until 28 days after last dose
Population: Safety Population: All treated participants. Additionally, 2 participants randomized to trastuzumab+taxane received 3 cycles of trastuzumab emtansine and were included in trastuzumab emtansine+placebo arm. 6 participants randomized to trastuzumab emtansine+placebo received pertuzumab and were included in trastuzumab emtansine+pertuzumab arm.
Measure: Number; unit: percentage of participants
Arm/Group | Trastuzumab + Taxane | Trastuzumab Emtansine + Placebo | Trastuzumab Emtansine + Pertuzumab
Number analyzed (Participants) | 353 | 361 | 366
percentage of participants | 54.1 | 45.4 | 46.2

11. Secondary Outcome: Percentage of Participants Who Died at 2 Years
Time Frame: From randomization until 2 years
Population: ITT Population
Measure: Number; unit: percentage of participants
Arm/Group | Trastuzumab + Taxane | Trastuzumab Emtansine + Placebo | Trastuzumab Emtansine + Pertuzumab
Number analyzed (Participants) | 365 | 367 | 363
percentage of participants | 20.3 | 20.2 | 19.6

12. Secondary Outcome: Overall Survival Truncated at 2 Years
Description: Overall Survival truncated at 2 years was defined as the percentage of participants alive at 2 years.
Time Frame: From randomization until 2 years
Population: ITT Population.
Measure: Number; unit: percentage of participants
Arm/Group | Trastuzumab + Taxane | Trastuzumab Emtansine + Placebo | Trastuzumab Emtansine + Pertuzumab
Number analyzed (Participants) | 365 | 367 | 363
percentage of participants | 79.7 [NA to NA] | 79.8 [NA to NA] | 80.4 [NA to NA]

13. Secondary Outcome: Percentage of Participants With Grade 5 Adverse Events
Description: Adverse events were graded according to NCI CTCAE version 4.0. Grade 5 adverse events are those events which led to death.
Time Frame: Up to 50 months from randomization until clinical cutoff of 16-Sept-2014 (continuously until 28 days after last dose)
Population: Safety population
Measure: Number; unit: percentage of participants
Arm/Group | Trastuzumab + Taxane | Trastuzumab Emtansine + Placebo | Trastuzumab Emtansine + Pertuzumab
Number analyzed (Participants) | 353 | 361 | 366
percentage of participants | 1.7 | 1.1 | 1.9

14. Secondary Outcome: Percentage of Participants With Grade 3-4 Laboratory Parameters
Description: Laboratory results were graded according to NCI CTCAE version 4.0. Grade 3: Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self care activity of daily living with inability to perform bathing, dressing and undressing, feeding self, using the toilet, taking medications but not bedridden. Grade 4: An immediate threat to life. Urgent medical intervention is required in order to maintain survival.
Time Frame: Day 1, 8, and 15 of Cycle 1-3 and on Day 1 of each subsequent cycle up to 50 months from randomization until clinical cutoff of 16-Sept-2014
Population: Safety population. Number of participants analyzed=participants with available data for the outcome.
Measure: Number; unit: percentage of participants
Arm/Group | Trastuzumab + Taxane | Trastuzumab Emtansine + Placebo | Trastuzumab Emtansine + Pertuzumab
Number analyzed (Participants) | 352 | 361 | 363
percentage of participants
  Hemoglobin-Low: Grade 3 | 4.3 | 5.8 | 6.9
  Neutrophils-Low: Grade 3 | 20.2 | 5.5 | 5.0
  Neutrophils-Low: Grade 4 | 43.8 | 1.9 | 0.8
  Platelets-Low: Grade 3 | 0.9 | 12.7 | 12.9
  Platelets-Low: Grade 4 | 0.3 | 2.8 | 2.5
  Alkaline Phosphate-High: Grade 3 | 1.1 | 3.9 | 3.0
  Alanine Transaminase-High: Grade 3 | 3.4 | 9.1 | 8.0
  Alanine Transaminase-High: Grade 4 | 0.0 | 0.3 | 0.6
  Aspartate Aminotransferase-High: Grade 3 | 1.1 | 11.9 | 6.9
  Aspartate Aminotransferase-High: Grade 4 | 0.0 | 0.3 | 0.3
  Creatinine-High: Grade 3 | 0.9 | 0.3 | 1.1
  Creatinine-High: Grade 4 | 0.0 | 0.0 | 0.3
  Potassium-Low: Grade 3 | 4.3 | 4.7 | 5.2
  Potassium-Low: Grade 4 | 0.6 | 1.7 | 0.6
  Total Bilirubin-High: Grade 3 | 0.3 | 0.3 | 0.3

15. Secondary Outcome: Percentage of Participants With Decline of ≥2 Points From Baseline in Eastern Cooperative Oncology Group (ECOG) Performance Status
Description: The ECOG performance status is a scale used to quantify cancer participants' general well-being and activities of daily life. The scale ranges from 0 to 5, with 0 denoting perfect health and 5 indicating death. The 6 categories are 0=Asymptomatic (Fully active, able to carry on all predisease activities without restriction), 1=Symptomatic but completely ambulatory (Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature), 2=Symptomatic, < 50% in bed during the day (Ambulatory and capable of all self-care but unable to carry out any work activities. Up and about more than 50% of waking hours), 3=Symptomatic, > 50% in bed, but not bedbound (Capable of only limited self-care, confined to bed or chair 50% or more of waking hours), 4=Bedbound (Completely disabled. Cannot carry on any self-care. Totally confined to bed or chair), 5=Death.
Time Frame: Baseline, Day 1 of every Cycle up to Clinical Data Cut (up to 48 months)
Population: Safety population
Measure: Number; unit: percentage of participants
Arm/Group | Trastuzumab + Taxane | Trastuzumab Emtansine + Placebo | Trastuzumab Emtansine + Pertuzumab
Number analyzed (Participants) | 353 | 361 | 366
percentage of participants | 7.6 | 6.1 | 7.9

16. Secondary Outcome: Hospitalization Days
Description: Hospitalization was defined as a non-administration-related hospitalization due to serious adverse event, while on study treatment. Reported values represent number of days admitted per participants.
Time Frame: Up to 48 months from randomization until clinical cutoff of 16-Sept-2014
Population: Safety population. Number of participants analyzed=participants with hospitalization and data available for calculation of the parameter.
Measure: Median (Full Range); unit: days
Arm/Group | Trastuzumab + Taxane | Trastuzumab Emtansine + Placebo | Trastuzumab Emtansine + Pertuzumab
Number analyzed (Participants) | 353 | 361 | 366
days | 6 [1 to 50] | 5 [1 to 117] | 8 [1 to 381]

17. Secondary Outcome: Percentage of Participants With Hospitalization
Description: Hospitalization was defined as a non-administration-related hospitalization due to serious adverse event, while on study treatment.
Time Frame: Up to 48 months from randomization until clinical cutoff of 16-Sept-2014
Population: Safety population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Trastuzumab + Taxane | Trastuzumab Emtansine + Placebo | Trastuzumab Emtansine + Pertuzumab
Number analyzed (Participants) | 353 | 361 | 366
percentage of participants | 21.8 [17.62 to 26.36] | 20.2 [16.20 to 24.71] | 22.1 [18.03 to 26.70]

18. Secondary Outcome: Percentage of Participants With Objective Response According to IRF Assessment
Description: Objective response was defined as having complete response (CR) or partial response (PR), assessed according to RECIST version 1.1, using radiographic images submitted to the IRF up to and including the confirmatory tumor assessment 4 to 6 weeks after study drug discontinuation. CR was defined as the disappearance of all target and non-target lesions and short-axis reduction in pathological lymph nodes to <10 mm. PR was defined as a ≥30% decrease in sum of diameters of target lesions, taking as reference the Baseline sum. Response was determined using 2 consecutive tumor assessments at least 4 weeks apart. The percentage of participants with a best overall response of CR or PR (ie, the objective response rate [ORR]) was calculated as [number of participants meeting the respective criteria divided by the number analyzed] multiplied by 100. Corresponding CIs were computed using the Blyth-Still-Casella exact method.
Time Frame: Up to 46 months from randomization until clinical cutoff of 16-Sept-2014 (at Screening, every 9 weeks for 81 weeks, then every 12 weeks thereafter and/or up to 42 days after last dose)
Population: ITT Population. Only participants with measurable disease at Baseline were included in the analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Trastuzumab + Taxane | Trastuzumab Emtansine + Placebo | Trastuzumab Emtansine + Pertuzumab
Number analyzed (Participants) | 287 | 303 | 299
percentage of participants | 67.9 [62.26 to 73.31] | 59.7 [54.07 to 65.30] | 64.2 [58.62 to 69.65]
Statistical Analysis 1: Comparison: Trastuzumab + Taxane vs Trastuzumab Emtansine + Placebo; Test type: Superiority or Other; Difference in Response Rate = -8.2, 95% CI 2-sided [-15.9 to -0.5] — Direction of comparison: Trastuzumab Emtansine + Placebo vs Trastuzumab + Taxane
Statistical Analysis 2: Comparison: Trastuzumab + Taxane vs Trastuzumab Emtansine + Pertuzumab; Test type: Superiority or Other; Difference in Response Rate = -3.7, 95% CI 2-sided [-11.4 to 3.9] — Direction of comparison: Trastuzumab Emtansine + Pertuzumab vs Trastuzumab + Taxane
Statistical Analysis 3: Comparison: Trastuzumab Emtansine + Placebo vs Trastuzumab Emtansine + Pertuzumab; Test type: Superiority or Other; Difference in Response Rate = 4.5, 95% CI 2-sided [-3.3 to 12.2] — Direction of comparison: Trastuzumab Emtansine + Pertuzumab vs Trastuzumab Emtansine + Placebo

19. Secondary Outcome: Percentage of Participants With Objective Response According to Investigator Assessment
Description: Objective response was defined as having CR or PR, assessed according to RECIST version 1.1, by investigator. CR was defined as the disappearance of all target and non-target lesions and short-axis reduction in pathological lymph nodes to <10 mm. PR was defined as a ≥30% decrease in sum of diameters of target lesions, taking as reference the Baseline sum. Response was determined using 2 consecutive tumor assessments at least 4 weeks apart. The percentage of participants with a best overall response of CR or PR (ie, the ORR) was calculated as [number of participants meeting the respective criteria divided by the number analyzed] multiplied by 100. Corresponding CIs were computed using the Blyth-Still-Casella exact method.
Time Frame: as for outcome 18
Population: ITT Population.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Trastuzumab + Taxane | Trastuzumab Emtansine + Placebo | Trastuzumab Emtansine + Pertuzumab
Number analyzed (Participants) | 365 | 367 | 363
percentage of participants | 69.3 [63.74 to 74.52] | 64.6 [59.12 to 69.87] | 67.5 [62.17 to 72.68]
Statistical Analysis 1: Comparison: Trastuzumab + Taxane vs Trastuzumab Emtansine + Placebo; Test type: Superiority or Other; Difference in Response Rate = -4.6, 95% CI 2-sided [-12.1 to 2.8] — Direction of comparison: Trastuzumab Emtansine + Placebo vs Trastuzumab + Taxane
Statistical Analysis 2: Comparison: Trastuzumab + Taxane vs Trastuzumab Emtansine + Pertuzumab; Test type: Superiority or Other; Difference in Response Rate = -1.8, 95% CI 2-sided [-9.2 to 5.7] — Direction of comparison: Trastuzumab Emtansine + Pertuzumab vs Trastuzumab + Taxane
Statistical Analysis 3: Comparison: Trastuzumab Emtansine + Placebo vs Trastuzumab Emtansine + Pertuzumab; Test type: Superiority or Other; Difference in Response Rate = 2.9, 95% CI 2-sided [-4.5 to 10.3] — Direction of comparison: Trastuzumab Emtansine + Pertuzumab vs Trastuzumab Emtansine + Placebo

20. Secondary Outcome: Duration of Response According to IRF Assessment
Description: Tumor assessments were performed according to RECIST version 1.1, using radiographic images submitted to the IRF up to and including the confirmatory tumor assessment 4 to 6 weeks after study drug discontinuation. Duration of response was defined as the time from confirmed PR or CR to first documented disease progression or death from any cause. CR was defined as the disappearance of all target lesions and non-target lesions and short-axis reduction in pathological lymph nodes to <10 mm. PR was defined as a ≥30% decrease in sum of diameters of target lesions, taking as reference the Baseline sum. Response was determined using 2 consecutive tumor assessments at least 4 weeks apart. Median duration of response was estimated using Kaplan-Meier analysis, and corresponding CIs were computed using the Brookmeyer-Crowley method.
Time Frame: as for outcome 18
Population: ITT Population. Only participants achieving CR or PR were included in the analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Trastuzumab + Taxane | Trastuzumab Emtansine + Placebo | Trastuzumab Emtansine + Pertuzumab
Number analyzed (Participants) | 195 | 181 | 192
months | 12.5 [10.5 to 16.6] | 20.7 [14.8 to 25.0] | 21.2 [15.8 to 29.3]
Statistical Analysis 1: Comparison: Trastuzumab + Taxane vs Trastuzumab Emtansine + Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; Hazard Ratio (HR) = 0.60, 97.5% CI 2-sided [0.43 to 0.84] — Direction of comparison: Trastuzumab Emtansine + Placebo vs Trastuzumab + Taxane
Statistical Analysis 2: Comparison: Trastuzumab + Taxane vs Trastuzumab Emtansine + Pertuzumab; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; Hazard Ratio (HR) = 0.62, 97.5% CI 2-sided [0.45 to 0.85] — Direction of comparison: Trastuzumab Emtansine + Pertuzumab vs Trastuzumab + Taxane

21. Secondary Outcome: Percentage of Participants With a Best Overall Response of CR, PR, or Stable Disease (SD) According to IRF Assessment
Description: Tumor assessments were performed according to RECIST version 1.1, using radiographic images submitted to the IRF up to and including the confirmatory tumor assessment 4 to 6 weeks after study drug discontinuation. CR was defined as the disappearance of all target and non-target lesions and short-axis reduction in pathological lymph nodes to <10 mm. PR was defined as a ≥30% decrease in sum of diameters of target lesions, taking as reference the Baseline sum. SD was defined as neither sufficient shrinkage to quality for PR nor sufficient (20%) increase to qualify for disease progression. Response was determined using 2 consecutive tumor assessments at least 4 weeks apart. The percentage of participants with a best overall response of CR, PR, or SD was calculated as [number of participants meeting the respective criteria divided by the number analyzed] multiplied by 100.
Time Frame: as for outcome 18
Population: Data were not analyzed. Protocol Amendment E removed this outcome measure as a secondary endpoint, because it was redundant to another prespecified secondary endpoint.
Arm/Group | Trastuzumab + Taxane | Trastuzumab Emtansine + Placebo | Trastuzumab Emtansine + Pertuzumab
Number analyzed (Participants) | 0 | 0 | 0

22. Secondary Outcome: Percentage of Participants Experiencing a Clinically Significant Increase in Taxane-Related Treatment Symptoms as Measured by Taxane Subscale of the Functional Assessment of Cancer Therapy (FACT) Taxane (FACT-TaxS) Score
Description: The FACT-Taxane is a self-reported instrument which measures the health-related quality of life (HRQOL) of participants receiving taxane-containing chemotherapy. The FACT-TaxS consists of 16 items including 11 neurotoxicity-related questions and 5 additional questions assessing arthralgia, myalgia, and skin discoloration. Items are rated from 0 (not at all) to 4 (very much) and a total score is inversely derived. Scores may range from 0 to 64, with higher scores indicating fewer/no symptoms. A minimally clinically important difference in treatment-related symptoms was defined as a ≥5% decrease (ie, 3.2 points) in FACT-TaxS score from Baseline. The percentage of participants with treatment-related symptoms was calculated using following formula: [number of participants meeting the above threshold divided by the number analyzed] multiplied by 100. Corresponding CIs were computed using the Blyth-Still-Casella exact method.
Time Frame: Up to 39 months from randomization until clinical cutoff of 16-Sept-2014 (at Baseline, on Day 1 of Cycles 2 to 8 and every even-numbered cycle thereafter and/or up to 42 days after last dose)
Population: ITT Population (Protocol Amendment C Subpopulation): All randomized participants who entered the study after Protocol Amendment C.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Trastuzumab + Taxane | Trastuzumab Emtansine + Placebo | Trastuzumab Emtansine + Pertuzumab
Number analyzed (Participants) | 173 | 171 | 154
percentage of participants | 93.1 [88.48 to 96.06] | 60.8 [53.39 to 67.93] | 68.8 [61.32 to 75.92]
Statistical Analysis 1: Comparison: Trastuzumab + Taxane vs Trastuzumab Emtansine + Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; Difference in Symptom Rate = -32.2, 95% CI 2-sided [-40 to -24] — Direction of comparison: Trastuzumab Emtansine + Placebo vs Trastuzumab + Taxane
Statistical Analysis 2: Comparison: Trastuzumab + Taxane vs Trastuzumab Emtansine + Pertuzumab; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; Difference in Symptom Rate = -24.2, 95% CI 2-sided [-32 to -16] — Direction of comparison: Trastuzumab Emtansine + Pertuzumab vs Trastuzumab + Taxane
Statistical Analysis 3: Comparison: Trastuzumab Emtansine + Placebo vs Trastuzumab Emtansine + Pertuzumab; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; Difference in Symptom Rate = 8.0, 95% CI 2-sided [-2.3 to 18.4] — Direction of comparison: Trastuzumab Emtansine + Pertuzumab vs Trastuzumab Emtansine + Placebo

23. Secondary Outcome: Percentage of Participants Reporting Nausea According to the Relevant Single Items of The FACT Colorectal Cancel (FACT-C) Module
Description: The FACT-C is a self-reported instrument which measures HRQOL pertaining to colorectal cancer. Response options on each question may range from 0 (not at all) to 4 (very much). The percentage of participants with nausea was calculated using following formula: [number of participants with any level of either symptom divided by the number analyzed] multiplied by 100.
Time Frame: At Baseline, Day 8 of Cycle 1, and Days 1 and 8 of Cycle 2
Population: ITT Population (Protocol Amendment C Subpopulation). Only participants with a FACT-C score at the designated visit (n) were included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Trastuzumab + Taxane | Trastuzumab Emtansine + Placebo | Trastuzumab Emtansine + Pertuzumab
Number analyzed (Participants) | 173 | 171 | 154
percentage of participants
  Nausea, Baseline (n=166,166,150) | 22.3 | 14.5 | 21.3
  Nausea, Cycle 1 Day 8 (n=121,114,95) | 38.0 | 36.0 | 52.6
  Nausea, Cycle 2 Day 1 (n=147,151,138) | 27.2 | 20.5 | 36.2
  Nausea, Cycle 2 Day 8 (n=122,121,105) | 35.2 | 28.1 | 45.7

24. Secondary Outcome: Percentage of Participants Reporting Diarrhea According to the Relevant Single Items of The FACT-C Module
Description: The FACT-C is a self-reported instrument which measures HRQOL pertaining to colorectal cancer. Response options on each question may range from 0 (not at all) to 4 (very much). The percentage of participants with diarrhea was calculated using following formula: [number of participants with any level of either symptom divided by the number analyzed] multiplied by 100.
Time Frame: At Baseline, Day 8 of Cycle 1, and Days 1 and 8 of Cycle 2
Population: as for outcome 23
Measure: Number; unit: percentage of participants
Arm/Group | Trastuzumab + Taxane | Trastuzumab Emtansine + Placebo | Trastuzumab Emtansine + Pertuzumab
Number analyzed (Participants) | 173 | 171 | 154
percentage of participants
  Diarrhea, Baseline (n=173,170,153) | 15.0 | 7.6 | 11.8
  Diarrhea, Cycle 1 Day 8 (n=124,117,98) | 34.7 | 17.9 | 34.7
  Diarrhea, Cycle 2 Day 1 (n=161,160,144) | 24.2 | 11.3 | 39.6
  Diarrhea, Cycle 2 Day 8 (n=125,123,107) | 34.4 | 8.1 | 41.1

25. Secondary Outcome: Percentage of Participants With a Clinically Significant Deterioration in Health Related Quality of Life (HRQoL) as Measured by FACT Breast (FACT-B) Trial Outcome Index-Physical Function Breast (TOI-PFB) Score
Description: The FACT-B is a self-reported instrument which measures HRQOL of participants with breast cancer. It consists of 5 subscales including physical well-being (PWB), social well-being (SWB), emotional well-being (EWB), functional well-being (FWB), and a breast cancer subscale (BCS). The TOI-PFB score is taken by adding the scores from the PWB (7 items), FWB (7 items), and BCS (9 items) subscales. Items are rated from 0 (not at all) to 4 (very much) and a total score is derived. Scores may range from 0 to 92, with higher scores indicating better HRQOL. A 5 point change has been identified as the clinically minimal important difference (CMID) on the FACT-TOI-PFB scale. The percentage of participants with deterioration was calculated as [number of participants meeting the above threshold divided by the number analyzed] multiplied by 100.
Time Frame: as for outcome 22
Population: ITT Population. Number of participants analyzed=participants with baseline and at least one post baseline FACT-B TOI-PFB score.
Measure: Number; unit: percentage of participants
Arm/Group | Trastuzumab + Taxane | Trastuzumab Emtansine + Placebo | Trastuzumab Emtansine + Pertuzumab
Number analyzed (Participants) | 327 | 352 | 338
percentage of participants | 61.8 | 50.9 | 50.6

26. Secondary Outcome: Time to Deterioration in HRQoL as Assessed by FACT-B TOI-PFB Score
Description: The FACT-B is a self-reported instrument which measures HRQOL of participants with breast cancer. It consists of 5 subscales including PWB, SWB, EWB, FWB, and BCS. The TOI-PFB score is taken by adding the scores from the PWB (7 items), FWB (7 items), and BCS (9 items) subscales. Items are rated from 0 (not at all) to 4 (very much) and a total score is derived. Scores may range from 0 to 92, with higher scores indicating better HRQOL. A 5 point change has been identified as the clinically minimal important difference (CMID) on the FACT-TOI-PFB scale. Time to deterioration was defined as the time from Baseline until the first decrease in FACT-B TOI-PFB score. Median time to deterioration was estimated using Kaplan-Meier analysis, and corresponding CIs were computed using the Brookmeyer-Crowley method.
Time Frame: Baseline up to 39 months from randomization until clinical cutoff of 16-Sept-2014
Population: as for outcome 25
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Trastuzumab + Taxane | Trastuzumab Emtansine + Placebo | Trastuzumab Emtansine + Pertuzumab
Number analyzed (Participants) | 327 | 352 | 338
months | 3.6 [3.0 to 4.4] | 7.7 [6.2 to 11.9] | 9.0 [5.1 to 14.5]
Statistical Analysis 1: Comparison: Trastuzumab + Taxane vs Trastuzumab Emtansine + Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; Hazard Ratio (HR) = 0.70, 95% CI 2-sided [0.57 to 0.86] — Direction of comparison: Trastuzumab Emtansine + Placebo vs Trastuzumab + Taxane
Statistical Analysis 2: Comparison: Trastuzumab + Taxane vs Trastuzumab Emtansine + Pertuzumab; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; Hazard Ratio (HR) = 0.68, 95% CI 2-sided [0.55 to 0.84] — Direction of comparison: Trastuzumab Emtansine + Pertuzumab vs Trastuzumab + Taxane

27. Secondary Outcome: Change From Baseline in Rotterdam Symptom Checklist (RSCL) Activity Level Scale Score
Description: The RSCL is a self-reported instrument which consists of 4 domains including physical symptom distress, psychological distress, activity level, and overall global life quality. Only the activity level scale was collected and assessed. Scores may range from 0 to 100, with higher scores indicating increased burden of disease. Mean RSCL activity scale score changes were calculated as [mean score at the assessment visit minus mean score at Baseline]. The higher the score, the higher the level of impairment or burden.
Time Frame: Baseline, Cycle 7 (Week 18)
Population: ITT Population. Here, 'n' signifies the number of participants with available data at baseline and Cycle 7 (Week 18).
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Trastuzumab + Taxane | Trastuzumab Emtansine + Placebo | Trastuzumab Emtansine + Pertuzumab
Number analyzed (Participants) | 365 | 367 | 363
units on a scale
  Baseline (n=344,355,344) | 85.0 [82.9 to 87.2] | 85.5 [83.3 to 87.8] | 85.7 [83.5 to 87.8]
  Change From Baseline at Cycle 7 (n=261,252,261) | -1.6 [-4.2 to 1.0] | 2.3 [0.4 to 4.2] | -0.2 [-2.1 to 1.6]

28. Secondary Outcome: Change From Baseline in Work Productivity According to Work Productivity and Activity Impairment (WPAI) Questionnaire Score
Description: The WPAI is a patient-reported measure which assesses the effect of general health and symptom severity on work productivity and regular activities. The General Health questionnaire asks participants to estimate the number of hours missed from work due to reasons related and unrelated to their health problems, as well as the total number of hours actually worked in the preceding 7-day period. The percentage of participants reporting that they were employed (working for pay) was assessed at baseline was assessed along with Absenteeism (work time missed), Presenteeism (impairment at work / reduced on-the-job effectiveness), Work productivity loss (overall work impairment / absenteeism plus presenteeism), and Activity Impairment. The reported changes represent change from baseline at Cycle 7. The score range for the scales of the WPAI is between 0 (no effect) to 100% (max effect)
Time Frame: Baseline, Cycle 7 (Week 18)
Population: Number of participants analysed=participants from ITT population who were employed at baseline. Here, 'n' signifies the number of participants with available data at specified category.
Measure: Mean (95% Confidence Interval); unit: percent of work
Arm/Group | Trastuzumab + Taxane | Trastuzumab Emtansine + Placebo | Trastuzumab Emtansine + Pertuzumab
Number analyzed (Participants) | 67 | 64 | 67
percent of work
  % Work Time Missed at Baseline (n=66,63,67) | 15.3 [9.2 to 21.4] | 9.5 [4.2 to 14.8] | 13.6 [7.7 to 19.6]
  Change in % Work Time Missed (n=35,33,36) | 0.4 [-7.3 to 8.2] | -0.0 [-4.5 to 4.5] | -4.3 [-13.0 to 4.6]
  % Impairment While Working at Baseline(n=67,64,67) | 20.0 [14.1 to 25.9] | 15.3 [9.5 to 21.1] | 19.9 [13.6 to 26.1]
  Change in % Impairment While Working (n=34,32,35) | 8.8 [2.0 to 15.6] | -0.3 [-11.0 to 10.5] | -2.7 [-11.0 to 5.2]
  % Overall Work Impairment at Baseline (n=65,62,66) | 28.5 [20.7 to 36.2] | 21.2 [13.8 to 28.7] | 28.1 [20.3 to 35.9]
  Change in % Overall Work Impairment (n=34,31,35) | 9.1 [-0.4 to 18.6] | -1.1 [-13.0 to 11.0] | -4.6 [-14.0 to 5.0]

29. Secondary Outcome: Change From Baseline in Activity Impairment According to Work Productivity and Activity Impairment (WPAI) Questionnaire Score
Description: as for outcome 28
Time Frame: Baseline, Cycle 7 (Week 18)
Population: Number of participants analysed=participants from ITT population who reported conduct of daily activities. Here, 'n' signifies the number of participants with available data at specified category.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Trastuzumab + Taxane | Trastuzumab Emtansine + Placebo | Trastuzumab Emtansine + Pertuzumab
Number analyzed (Participants) | 312 | 334 | 321
units on a scale
  % Activity Impairment at Baseline (n=312,334,321) | 32.9 [29.6 to 36.3] | 33.6 [30.2 to 37.0] | 32.7 [29.5 to 36.0]
  Change in % Activity Impairment (n=227,222,234) | 4.5 [0.2 to 8.7] | -5.3 [-9.5 to -1.1] | -3.7 [-7.2 to -0.1]

30. Secondary Outcome: Percentage of Participants With a Best Overall Response of CR or PR According to IRF Assessment Among Those With High Human Epidermal Growth Factor Receptor 2 (HER2) Messenger Ribonucleic Acid (mRNA) Levels
Description: Tumor assessments were performed according to RECIST version 1.1, using radiographic images submitted to the IRF up to and including the confirmatory tumor assessment 4 to 6 weeks after study drug discontinuation. CR was defined as the disappearance of all target and non-target lesions and short-axis reduction in pathological lymph nodes to <10 mm. PR was defined as a ≥30% decrease in sum of diameters of target lesions, taking as reference the Baseline sum. Response was determined using 2 consecutive tumor assessments at least 4 weeks apart. The percentage of participants with a best overall response of CR or PR (ie, the ORR) was calculated as [number of participants meeting the respective criteria divided by the number analyzed] multiplied by 100.
Time Frame: as for outcome 18
Population: ITT Population (High HER2 mRNA Subpopulation): All randomized participants with above-the-median HER2 mRNA expression (value greater than [>] 59.71). Only participants with measurable disease at Baseline were included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Trastuzumab + Taxane | Trastuzumab Emtansine + Placebo | Trastuzumab Emtansine + Pertuzumab
Number analyzed (Participants) | 132 | 136 | 147
percentage of participants | 75.0 | 66.9 | 63.9
Statistical Analysis 1: Comparison: Trastuzumab + Taxane vs Trastuzumab Emtansine + Placebo; Test type: Superiority or Other; Odds Ratio (OR) = 0.67, 95% CI 2-sided [0.40 to 1.15] — Direction of comparison: Trastuzumab Emtansine + Placebo vs Trastuzumab + Taxane

31. Secondary Outcome: Percentage of Participants With a Best Overall Response of CR or PR According to IRF Assessment Among Those With Low HER2 mRNA Levels
Description: as for outcome 30
Time Frame: as for outcome 18
Population: ITT Population (Low HER2 mRNA Subpopulation): All randomized participants with below-the-median HER2 mRNA expression (value less than or equal to [≤] 59.71). Only participants with measurable disease at Baseline were included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Trastuzumab + Taxane | Trastuzumab Emtansine + Placebo | Trastuzumab Emtansine + Pertuzumab
Number analyzed (Participants) | 126 | 147 | 127
percentage of participants | 61.9 | 51.7 | 66.1
Statistical Analysis 1: Comparison: Trastuzumab + Taxane vs Trastuzumab Emtansine + Placebo; Test type: Superiority or Other; Odds Ratio (OR) = 0.66, 95% CI 2-sided [0.41 to 1.07] — Direction of comparison: Trastuzumab Emtansine + Placebo vs Trastuzumab + Taxane

32. Secondary Outcome: Percentage of Participants With Death or Disease Progression According to IRF Assessment Among Those With High HER2 mRNA Levels
Description: Tumor assessments were performed according to RECIST version 1.1, using radiographic images submitted to the IRF up to and including the confirmatory tumor assessment 4 to 6 weeks after study drug discontinuation. Disease progression was defined as a ≥20% and 5-mm increase in sum of diameters of target lesions, taking as reference the smallest sum obtained during the study, or appearance of new lesion(s). The percentage of participants with death or disease progression was calculated as [number of participants with event divided by the number analyzed] multiplied by 100.
Time Frame: as for outcome 1
Population: ITT Population (High HER2 mRNA Subpopulation).
Measure: Number; unit: percentage of participants
Arm/Group | Trastuzumab + Taxane | Trastuzumab Emtansine + Placebo | Trastuzumab Emtansine + Pertuzumab
Number analyzed (Participants) | 160 | 165 | 173
percentage of participants | 59.4 | 57.6 | 56.1

33. Secondary Outcome: PFS According to IRF Assessment Among Those With High HER2 mRNA Levels
Description: Tumor assessments were performed according to RECIST version 1.1, using radiographic images submitted to the IRF up to and including the confirmatory tumor assessment 4 to 6 weeks after study drug discontinuation. PFS was defined as the time from randomization to first documented disease progression or death from any cause. Disease progression was defined as a ≥20% and 5-mm increase in sum of diameters of target lesions, taking as reference the smallest sum obtained during the study, or appearance of new lesion(s). Median duration of PFS was estimated using Kaplan-Meier analysis.
Time Frame: as for outcome 1
Population: ITT Population (High HER2 mRNA Subpopulation).
Measure: Median (Full Range); unit: months
Arm/Group | Trastuzumab + Taxane | Trastuzumab Emtansine + Placebo | Trastuzumab Emtansine + Pertuzumab
Number analyzed (Participants) | 160 | 165 | 173
months | 15.9 [0.1 to 46.4] | 18.6 [0.1 to 46.0] | 18.7 [0.1 to 48.1]
Statistical Analysis 1: Comparison: Trastuzumab + Taxane vs Trastuzumab Emtansine + Placebo; Test type: Superiority or Other; Hazard Ratio (HR) = 0.90, 97.5% CI 2-sided [0.65 to 1.25] — Direction of comparison: Trastuzumab Emtansine + Placebo vs Trastuzumab + Taxane

34. Secondary Outcome: Percentage of Participants With Death or Disease Progression According to IRF Assessment Among Those With Low HER2 mRNA Levels
Description: as for outcome 32
Time Frame: as for outcome 1
Population: ITT Population (Low HER2 mRNA Subpopulation).
Measure: Number; unit: percentage of participants
Arm/Group | Trastuzumab + Taxane | Trastuzumab Emtansine + Placebo | Trastuzumab Emtansine + Pertuzumab
Number analyzed (Participants) | 170 | 174 | 157
percentage of participants | 66.5 | 70.1 | 62.4

35. Secondary Outcome: PFS According to IRF Assessment Among Those With Low HER2 mRNA Levels
Description: as for outcome 33
Time Frame: as for outcome 1
Population: ITT Population (Low HER2 mRNA Subpopulation).
Measure: Median (Full Range); unit: months
Arm/Group | Trastuzumab + Taxane | Trastuzumab Emtansine + Placebo | Trastuzumab Emtansine + Pertuzumab
Number analyzed (Participants) | 170 | 174 | 157
months | 12.4 [0.1 to 47.3] | 10.2 [0.1 to 43.6] | 14.5 [0.1 to 40.7]
Statistical Analysis 1: Comparison: Trastuzumab + Taxane vs Trastuzumab Emtansine + Placebo; Test type: Superiority or Other; Hazard Ratio (HR) = 1.00, 97.5% CI 2-sided [0.74 to 1.34] — Direction of comparison: Trastuzumab Emtansine + Placebo vs Trastuzumab + Taxane

36. Secondary Outcome: Percentage of Participants Who Died Prior to Clinical Cutoff Among Those With High HER2 mRNA Levels
Description: as for outcome 3
Time Frame: as for outcome 3
Population: ITT Population (High HER2 mRNA Subpopulation).
Measure: Number; unit: percentage of participants
Arm/Group | Trastuzumab + Taxane | Trastuzumab Emtansine + Placebo | Trastuzumab Emtansine + Pertuzumab
Number analyzed (Participants) | 160 | 165 | 173
percentage of participants | 38.8 | 41.2 | 45.1

37. Secondary Outcome: OS at Clinical Cutoff Among Those With High HER2 mRNA Levels
Description: OS was defined as the time from randomization to death from any cause. Median duration of OS was estimated using Kaplan-Meier analysis.
Time Frame: as for outcome 3
Population: ITT Population (High HER2 mRNA Subpopulation).
Measure: Median (Full Range); unit: months
Arm/Group | Trastuzumab + Taxane | Trastuzumab Emtansine + Placebo | Trastuzumab Emtansine + Pertuzumab
Number analyzed (Participants) | 160 | 165 | 173
months | NA [50.86 to NA] — Median duration of OS was not reached due to insufficient follow-up. Upper limit of CI was not reached due to low number of participants with events. | 65.97 [54.54 to 67.98] | 55.39 [48.23 to NA] — Upper limit of CI was not reached due to low number of participants with events.

38. Secondary Outcome: Percentage of Participants Who Died Prior to Clinical Cutoff Among Those With Low HER2 mRNA Levels
Description: as for outcome 3
Time Frame: as for outcome 3
Population: ITT Population (Low HER2 mRNA Subpopulation).
Measure: Number; unit: percentage of participants
Arm/Group | Trastuzumab + Taxane | Trastuzumab Emtansine + Placebo | Trastuzumab Emtansine + Pertuzumab
Number analyzed (Participants) | 170 | 174 | 157
percentage of participants | 51.8 | 52.9 | 45.2

39. Secondary Outcome: OS at Clinical Cutoff Among Those With Low HER2 mRNA Levels
Description: OS was defined as the time from randomization to death from any cause. Median duration of OS was estimated using Kaplan-Meier analysis. Reported upper bound of confidence interval for "Trastuzumab Emtansine + Placebo" and confidence interval values for "Trastuzumab + Taxane" and "Trastuzumab Emtansine + Pertuzumab" are censored values.
Time Frame: as for outcome 3
Population: ITT Population (Low HER2 mRNA Subpopulation).
Measure: Median (Full Range); unit: months
Arm/Group | Trastuzumab + Taxane | Trastuzumab Emtansine + Placebo | Trastuzumab Emtansine + Pertuzumab
Number analyzed (Participants) | 170 | 174 | 157
months | 43.96 [37.19 to 54.87] | 47.84 [42.09 to 53.85] | 53.29 [46.75 to NA] — Upper limit of CI was not reached due to low number of participants with events.

ADVERSE EVENTS:
Time Frame: Up to 70 months from randomization until clinical cutoff of 16 September 2016 (every 3 months until death, loss to follow-up, withdrawal, or study termination).
Description: Safety Population: All randomized participants who received at least one dose of study treatment and the participants were analyzed based on the treatment they actually received (N=353 in Trastuzumab + Taxane arm, N=361 in Trastuzumab Emtansine, Pertuzumab-placebo arm, N=366 in Trastuzumab emtansine + pertuzumab arm).
Arm/Group | Trastuzumab + Taxane | Trastuzumab Emtansine + Placebo | Trastuzumab Emtansine + Pertuzumab
Serious Adverse Events (participants affected / at risk) | 81/353 | 86/361 | 93/366
Other Adverse Events (participants affected / at risk) | 342/353 | 352/361 | 352/366
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Trastuzumab + Taxane (N=353) | Trastuzumab Emtansine + Placebo (N=361) | Trastuzumab Emtansine + Pertuzumab (N=366)
Febrile neutropenia (Blood and lymphatic system disorders) | 13 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 1 | 5 | 6
Neutropenia (Blood and lymphatic system disorders) | 5 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 2 | 2
Hypercoagulation (Blood and lymphatic system disorders) | 1 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 1
Cardiac failure (Cardiac disorders) | 0 | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 1
Myocardial infarction (Cardiac disorders) | 1 | 0 | 0
Pericardial effusion (Cardiac disorders) | 1 | 0 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 1
Ventricular tachycardia (Cardiac disorders) | 0 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 2
Blindness transient (Eye disorders) | 0 | 1 | 0
Macular hole (Eye disorders) | 0 | 1 | 0
Ocular hypertension (Eye disorders) | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 4 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 4
Abdominal pain (Gastrointestinal disorders) | 2 | 1 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 2
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Anal fistula (Gastrointestinal disorders) | 0 | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 0 | 1
Diverticulum (Gastrointestinal disorders) | 1 | 0 | 0
Gastric haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Gastric ulcer (Gastrointestinal disorders) | 0 | 1 | 0
Gastritis erosive (Gastrointestinal disorders) | 1 | 0 | 0
Large intestine perforation (Gastrointestinal disorders) | 1 | 0 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Mallory-Weiss syndrome (Gastrointestinal disorders) | 0 | 0 | 1
Mouth haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 1
Splenic artery aneurysm (Gastrointestinal disorders) | 0 | 1 | 0
Umbilical hernia (Gastrointestinal disorders) | 0 | 0 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Pyrexia (General disorders) | 2 | 4 | 5
Fatigue (General disorders) | 3 | 1 | 1
Non-cardiac chest pain (General disorders) | 0 | 2 | 1
Death (General disorders) | 0 | 1 | 0
General physical health deterioration (General disorders) | 0 | 0 | 2
Pain (General disorders) | 0 | 0 | 2
Asthenia (General disorders) | 0 | 0 | 1
Catheter site haematoma (General disorders) | 0 | 0 | 1
Malaise (General disorders) | 0 | 0 | 1
Oedema (General disorders) | 1 | 0 | 0
Peripheral swelling (General disorders) | 1 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 1 | 1
Hypersensitivity (Immune system disorders) | 0 | 2 | 2
Anaphylactic reaction (Immune system disorders) | 2 | 0 | 1
Cytokine release syndrome (Immune system disorders) | 0 | 0 | 1
Pneumonia (Infections and infestations) | 4 | 3 | 5
Cellulitis (Infections and infestations) | 3 | 3 | 1
Sepsis (Infections and infestations) | 1 | 0 | 4
Device related infection (Infections and infestations) | 0 | 1 | 1
Gastroenteritis (Infections and infestations) | 1 | 0 | 2
Infection (Infections and infestations) | 1 | 1 | 1
Neutropenic sepsis (Infections and infestations) | 3 | 0 | 0
Septic shock (Infections and infestations) | 2 | 1 | 1
Bronchitis (Infections and infestations) | 0 | 0 | 3
Herpes zoster (Infections and infestations) | 2 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 1 | 0
Urinary tract infection (Infections and infestations) | 2 | 0 | 0
Wound infection (Infections and infestations) | 1 | 1 | 0
Arthritis infective (Infections and infestations) | 0 | 1 | 0
Atypical pneumonia (Infections and infestations) | 0 | 0 | 1
Breast abscess (Infections and infestations) | 0 | 1 | 0
Chorioretinitis (Infections and infestations) | 0 | 0 | 1
Clostridium difficile colitis (Infections and infestations) | 0 | 0 | 1
Clostridium difficile infection (Infections and infestations) | 0 | 0 | 1
Cystitis (Infections and infestations) | 1 | 0 | 0
Empyema (Infections and infestations) | 0 | 0 | 1
Erysipelas (Infections and infestations) | 1 | 1 | 0
Escherichia sepsis (Infections and infestations) | 1 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 1
Influenza (Infections and infestations) | 1 | 1 | 0
Klebsiella sepsis (Infections and infestations) | 0 | 1 | 0
Localised infection (Infections and infestations) | 0 | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 0 | 1 | 0
Lung infection (Infections and infestations) | 1 | 0 | 0
Mastitis (Infections and infestations) | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0 | 0
Pneumonia pneumococcal (Infections and infestations) | 1 | 0 | 0
Rectal abscess (Infections and infestations) | 0 | 0 | 1
Respiratory tract infection (Infections and infestations) | 0 | 0 | 1
Streptococcal sepsis (Infections and infestations) | 1 | 0 | 0
Tooth infection (Infections and infestations) | 0 | 0 | 1
Urosepsis (Infections and infestations) | 1 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 7 | 13
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0 | 3
Pubis fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Arterial injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 2 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Gastrointestinal stoma complication (Injury, poisoning and procedural complications) | 1 | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Radiation retinopathy (Injury, poisoning and procedural complications) | 0 | 1 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 1
Wound secretion (Injury, poisoning and procedural complications) | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 2
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 2
Body temperature increased (Investigations) | 0 | 1 | 0
International normalised ratio increased (Investigations) | 1 | 0 | 0
Oxygen saturation decreased (Investigations) | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 2 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 2 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Exostosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Acute leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Chronic myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Colon neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Squamous cell carcinoma of the cervix (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 2 | 2
Syncope (Nervous system disorders) | 0 | 2 | 1
Haemorrhage intracranial (Nervous system disorders) | 1 | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 1
Cognitive disorder (Nervous system disorders) | 1 | 0 | 0
Depressed level of consciousness (Nervous system disorders) | 1 | 0 | 0
Guillain-Barre syndrome (Nervous system disorders) | 0 | 0 | 1
Lacunar infarction (Nervous system disorders) | 1 | 0 | 0
Paraparesis (Nervous system disorders) | 0 | 0 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 1 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 1
Vascular dementia (Nervous system disorders) | 0 | 1 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 2
Depression (Psychiatric disorders) | 0 | 1 | 2
Anxiety (Psychiatric disorders) | 0 | 0 | 1
Calculus urinary (Renal and urinary disorders) | 1 | 0 | 0
Menorrhagia (Reproductive system and breast disorders) | 0 | 1 | 1
Endometrial hypertrophy (Reproductive system and breast disorders) | 0 | 0 | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 3
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 4 | 2 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 3
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Alveolitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Nasal turbinate hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 2 | 0
Dermatomyositis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Peau d'orange (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Hypertension (Vascular disorders) | 1 | 1 | 0
Haematoma (Vascular disorders) | 0 | 2 | 0
Haemorrhage (Vascular disorders) | 0 | 0 | 1
Hypertensive crisis (Vascular disorders) | 0 | 0 | 1
Hypotension (Vascular disorders) | 1 | 0 | 0
Acute Myocardial Infarction (Cardiac disorders) | 1 | 0 | 0
Abdominal Discomfort (Gastrointestinal disorders) | 0 | 0 | 1
Ascites (Gastrointestinal disorders) | 0 | 1 | 0
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Haemorrhoidal Haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Adverse Drug Reaction (General disorders) | 0 | 0 | 1
Sudden Death (General disorders) | 0 | 0 | 1
Hepatic Fibrosis (Hepatobiliary disorders) | 0 | 1 | 0
Anaphylactic Shock (Immune system disorders) | 0 | 1 | 0
Anaphylactoid Reaction (Immune system disorders) | 0 | 0 | 1
Abscess Limb (Infections and infestations) | 0 | 1 | 0
Appendicitis Perforated (Infections and infestations) | 0 | 1 | 0
Catheter Site Infection (Infections and infestations) | 0 | 0 | 1
Skin Infection (Infections and infestations) | 0 | 0 | 1
Abdominal Injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Foot Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Stomal Hernia (Injury, poisoning and procedural complications) | 1 | 0 | 0
Diabetes Mellitus (Metabolism and nutrition disorders) | 0 | 0 | 1
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Intracranial Tumour Haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Cerebral Haemorrhage (Nervous system disorders) | 0 | 0 | 1
Epilepsy (Nervous system disorders) | 0 | 1 | 0
Neuropathy Peripheral (Nervous system disorders) | 0 | 0 | 1
Sciatica (Nervous system disorders) | 1 | 0 | 1
Seizure (Nervous system disorders) | 1 | 1 | 1
Device Breakage (Product Issues) | 0 | 1 | 0
Mental Status Changes (Psychiatric disorders) | 0 | 0 | 1
Suicide Attempt (Psychiatric disorders) | 1 | 0 | 0
Acute Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Cutaneous Lupus Erythematosus (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Aneurysm (Vascular disorders) | 0 | 0 | 1
Hypovolaemic Shock (Vascular disorders) | 0 | 0 | 1
Orthostatic Hypotension (Vascular disorders) | 0 | 1 | 0
Hepatic Haematoma (Hepatobiliary disorders) | 0 | 0 | 1
Uncoded serious adverse event (Injury, poisoning and procedural complications) | 0 | 0 | 1 — Per investigator, this serious adverse event was, "gamma nail implant broke (status after femur fracture)."
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Trastuzumab + Taxane (N=353) | Trastuzumab Emtansine + Placebo (N=361) | Trastuzumab Emtansine + Pertuzumab (N=366)
Nausea (Gastrointestinal disorders) | 131 | 174 | 192
Diarrhoea (Gastrointestinal disorders) | 173 | 92 | 178
Fatigue (General disorders) | 128 | 120 | 130
Headache (Nervous system disorders) | 80 | 116 | 120
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 53 | 113 | 127
Pyrexia (General disorders) | 59 | 96 | 118
Alopecia (Skin and subcutaneous tissue disorders) | 212 | 26 | 33
Vomiting (Gastrointestinal disorders) | 69 | 80 | 111
Decreased appetite (Metabolism and nutrition disorders) | 76 | 84 | 84
Arthralgia (Musculoskeletal and connective tissue disorders) | 91 | 83 | 71
Rash (Skin and subcutaneous tissue disorders) | 86 | 62 | 89
Constipation (Gastrointestinal disorders) | 72 | 82 | 71
Cough (Respiratory, thoracic and mediastinal disorders) | 74 | 72 | 79
Neuropathy peripheral (Nervous system disorders) | 99 | 52 | 69
Myalgia (Musculoskeletal and connective tissue disorders) | 82 | 66 | 61
Asthenia (General disorders) | 57 | 62 | 63
Chills (General disorders) | 14 | 55 | 97
Upper respiratory tract infection (Infections and infestations) | 55 | 50 | 66
Oedema peripheral (General disorders) | 98 | 37 | 35
Peripheral sensory neuropathy (Nervous system disorders) | 70 | 47 | 46
Back pain (Musculoskeletal and connective tissue disorders) | 46 | 60 | 63
Nasopharyngitis (Infections and infestations) | 49 | 52 | 66
Insomnia (Psychiatric disorders) | 51 | 51 | 52
Neutropenia (Blood and lymphatic system disorders) | 74 | 44 | 37
Pain in extremity (Musculoskeletal and connective tissue disorders) | 48 | 53 | 54
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 56 | 42 | 53
Anaemia (Blood and lymphatic system disorders) | 39 | 48 | 59
Dysgeusia (Nervous system disorders) | 54 | 30 | 50
Stomatitis (Gastrointestinal disorders) | 57 | 37 | 42
Dyspepsia (Gastrointestinal disorders) | 38 | 33 | 48
Abdominal pain upper (Gastrointestinal disorders) | 31 | 39 | 46
Dry mouth (Gastrointestinal disorders) | 13 | 52 | 45
Mucosal inflammation (General disorders) | 40 | 29 | 36
Paraesthesia (Nervous system disorders) | 41 | 31 | 43
Pruritus (Skin and subcutaneous tissue disorders) | 32 | 28 | 51
Dizziness (Nervous system disorders) | 35 | 38 | 38
Abdominal pain (Gastrointestinal disorders) | 31 | 35 | 41
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 52 | 61
Hypertension (Vascular disorders) | 19 | 37 | 43
Muscle spasms (Musculoskeletal and connective tissue disorders) | 15 | 32 | 62
Urinary tract infection (Infections and infestations) | 29 | 31 | 41
Nail disorder (Skin and subcutaneous tissue disorders) | 39 | 11 | 19
Aspartate aminotransferase increased (Investigations) | 9 | 54 | 28
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 29 | 31 | 30
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 23 | 30 | 37
Alanine aminotranseferase increased (Investigations) | 10 | 41 | 35
Anxiety (Psychiatric disorders) | 22 | 26 | 33
Lacrimation increased (Eye disorders) | 48 | 13 | 19
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 26 | 21 | 32
Bone pain (Musculoskeletal and connective tissue disorders) | 33 | 17 | 29
Influenza like illness (General disorders) | 17 | 31 | 32
Non-cardiac chest pain (General disorders) | 24 | 25 | 27
Dry skin (Skin and subcutaneous tissue disorders) | 24 | 24 | 29
Pain (General disorders) | 29 | 26 | 19
Depression (Psychiatric disorders) | 17 | 34 | 20
Dry eye (Eye disorders) | 13 | 25 | 24
Gingival bleeding (Gastrointestinal disorders) | 4 | 31 | 25
Hypokalaemia (Metabolism and nutrition disorders) | 15 | 19 | 30
Rhinitis (Infections and infestations) | 18 | 25 | 24
Influenza (Infections and infestations) | 14 | 22 | 25
Paronychia (Infections and infestations) | 22 | 8 | 30
Weight decreased (Investigations) | 7 | 24 | 30
Erythema (Skin and subcutaneous tissue disorders) | 24 | 13 | 20
Pharyngitis (Infections and infestations) | 14 | 19 | 17
Ejection fraction decreased (Investigations) | 31 | 7 | 16
Hot flush (Vascular disorders) | 27 | 16 | 12
Conjunctivitis (Infections and infestations) | 21 | 14 | 17
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 17 | 13 | 20
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 6 | 16 | 27
Breast pain (Reproductive system and breast disorders) | 18 | 13 | 16
Neck Pain (Musculoskeletal and connective tissue disorders) | 12 | 12 | 24
Gamma- glutamyltranseferase increased (Investigations) | 1 | 30 | 17
Oedema (General disorders) | 31 | 11 | 3
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 26 | 6 | 11
Haemorrhoids (Gastrointestinal disorders) | 9 | 12 | 22
Lymphoedema (Vascular disorders) | 27 | 7 | 8
Nail discolouration (Skin and subcutaneous tissue disorders) | 25 | 5 | 1
Vision Blurred (Eye disorders) | 10 | 13 | 19
Bronchitis (Infections and infestations) | 14 | 9 | 20
Onychoclasis (Skin and subcutaneous tissue disorders) | 13 | 19 | 17
Vertigo (Ear and labyrinth disorders) | 11 | 17 | 21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.